CLINICAL TRIAL: NCT02929823
Title: A Double-Masked, Randomized, Multicenter, Placebo-Controlled, Parallel-Group Study of SJP-0035 Ophthalmic Solution Compared With Placebo to Assess Safety and Efficacy of Two Dose Concentrations of SJP-0035 Ophthalmic Solution for Corneal Epithelial Wound Healing in Patients With Moderate to Severe Corneal Epithelial Disorders
Brief Title: Safety and Efficacy of SJP-0035 Ophthalmic Solution in Patients With Moderate to Severe Corneal Epithelial Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Senju Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJP-0035/2-02
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2018-05

CONDITIONS: Corneal Epithelial Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose SJP-0035 Ophthalmic solution (Experimental): Patients will administer 1 drop of 0.0002% SJP-0035 ophthalmic solution in the affected eye(s) 4 times daily for 4 weeks.
  Interventions: Drug: Low Dose SJP-0035 Ophthalmic Solution
- High Dose SJP-0035 Ophthalmic solution (Experimental): Patients will administer 1 drop of 0.001% SJP-0035 ophthalmic solution in the affected eye(s) 4 times daily for 4 weeks.
  Interventions: Drug: High Dose SJP-0035 Ophthalmic Solution
- Vehicle of SJP-0035 Ophthalmic solution (Placebo Comparator): Patients will administer 1 drop of 0% SJP-0035 ophthalmic solution (consisting of the vehicle for the solution) in the affected eye(s) 4 times daily for 4 weeks
  Interventions: Drug: Vehicle of SJP-0035 Ophthalmic solution

INTERVENTIONS:
Drug: High Dose SJP-0035 Ophthalmic Solution — 0.001% SJP-0035 Ophthalmic Solution
  Arms: High Dose SJP-0035 Ophthalmic solution
Drug: Low Dose SJP-0035 Ophthalmic Solution — 0.0002% SJP-0035 Ophthalmic Solution
  Arms: Low Dose SJP-0035 Ophthalmic solution
Drug: Vehicle of SJP-0035 Ophthalmic solution — 0% SJP-0035 Ophthalmic Solution
  Other Names: Placebo
  Arms: Vehicle of SJP-0035 Ophthalmic solution

SUMMARY:
The purpose of this study is to determine whether SJP-0035 ophthalmic solution is effective in promoting corneal epithelial wound healing in conditions associated with corneal epithelial disorders.

DETAILED DESCRIPTION:
There are currently no approved products available anywhere worldwide for the treatment of corneal epithelial disorders that directly affect the epithelia.

A Phase 1 study, Study SJP-0035/1-01, was conducted in healthy volunteers to investigate the safety, tolerability, and pharmacokinetic profile of SJP-0035 ophthalmic solution, and to determine the appropriate dose to be evaluated in patients with moderate to severe corneal epithelial disorders. A Phase 2a study, Study SJP-0035/2-01, was conducted in patients with corneal epithelial disorders to evaluate the efficacy and safety of SJP-0035.

This Phase 2a study (Study SJP-0035/2-02) is being conducted to evaluate the safety and efficacy of 2 doses of SJP-0035 ophthalmic solution in patients with corneal epithelial disorders. The study will evaluate if SJP-0035 ophthalmic solution is able to promote corneal epithelial wound healing in patients with corneal epithelial disorders using 2 doses of SJP-0035 ophthalmic solution (0.0002% and 0.001%) that are lower than what was used in the previous Phase 2a study (Study SJP-0035/2-01; 0.005%).

ELIGIBILITY:
Inclusion Criteria:

* Is capable of understanding the written informed consent form (ICF), provides signed and witnessed written ICF, and agrees to comply with protocol requirements, including all required study visits
* Is a male or female 18 years of age or older
* Has a moderate to severe corneal epithelial disorder in both eyes
* Has blurred vision caused by corneal epithelial disorders in both eyes at Screening and Randomization
* Is a female of childbearing potential with a negative pregnancy test result at Screening and Randomization and agrees to use effective contraception throughout the study, or is a postmenopausal woman with a negative pregnancy test result at Screening and Randomization

Exclusion Criteria:

* Has any corneal stromal or endothelial abnormalities including an active bacterial or viral ocular infection, bullous keratopathy, chemical burns, or any trauma to the cornea in either eye at Screening and Randomization
* Has any active or chronic allergic, bacterial, or viral infection of ocular adnexa and eye structures in either eye at Screening and Randomization
* Has had intraocular surgery (including cataract or vitreous) in either eye within the last 30 days prior to the first dose of study drug
* Has had refractive surgery (including ocular surface laser surgery) in either eye within the last 6 months prior to the first dose of study drug
* Has used any ocular medication (except mydriatics, stain, and topical anesthesia used for study assessments) in either eye within 14 days prior to the first dose of study drug, or is anticipated to require such medications during the study.
* Is a contact lens wearer and cannot discontinue use in both eyes from Screening through EOS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Senju Investigational Site, Little Rock, Arkansas
  - Senju Investigational Site, Glendora, California
  - Senju Investigational Site, Lancaster, California
  - Senju Investigational Site, Long Beach, California
  - Senju Investigational Site, Montebello, California
  - Senju Investigational Site, Pasadena, California
  - Senju Investigational Site, Santa Ana, California
  - Senju Investigational Site, Miami, Florida
  - Senju Investigational Site, Hoffman Estates, Illinois
  - Senju Investigational Site, Edgewood, Kentucky
  - Senju Investigational Site, Louisville, Kentucky
  - Senju Investigational Site, Kansas City, Missouri
  - Senju Investigational Site, High Point, North Carolina
  - Senju Investigational Site, Rapid City, South Dakota
  - Senju Investigational Site, Cedar Park, Texas
  - Senju Investigational Site, Houston, Texas
  - Senju Investigational Site, Irving, Texas
  - Senju Investigational Site, Falls Church, Virginia
  - Senju Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at study sites in the USA and were assigned to study drug only if they met all the inclusion criteria and none of the exclusion criteria. Deviations from the inclusion/exclusion criteria were not permitted.
Pre-assignment Details: For patients using prohibited concomitant medications within 14 days prior to planned randomization date, a 14 day washout period was required prior to first dose of study drug. Patients who failed initial screening were allowed to rescreen once.
Groups:
- Placebo: Patients will administer 1 drop of 0% SJP-0035 ophthalmic solution (consisting of the vehicle for the solution) in the affected eye(s) 4 times daily for 4 weeks
  Vehicle of SJP-0035 Ophthalmic solution: 0% SJP-0035 Ophthalmic Solution
- 0.0002% SJP-0035 Ophthalmic Solution: Patients will administer 1 drop of 0.0002% SJP-0035 ophthalmic solution in the affected eye(s) 4 times daily for 4 weeks.
  Low Dose SJP-0035 Ophthalmic Solution: 0.0002% SJP-0035 Ophthalmic Solution
- 0.001% SJP-0035 Ophthalmic Solution: Patients will administer 1 drop of 0.001% SJP-0035 ophthalmic solution in the affected eye(s) 4 times daily for 4 weeks.
  High Dose SJP-0035 Ophthalmic Solution: 0.001% SJP-0035 Ophthalmic Solution
Period: Overall Study
Arm/Group | Placebo | 0.0002% SJP-0035 Ophthalmic Solution | 0.001% SJP-0035 Ophthalmic Solution
Started | 42 | 46 | 42
Completed | 39 | 40 | 38
Not Completed | 3 | 6 | 4

BASELINE CHARACTERISTICS:
Population: Safety Set: consisted of all participants who received any study drug. All analyses using the safety set grouped participants according to treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.0002% SJP-0035 Ophthalmic Solution | 0.001% SJP-0035 Ophthalmic Solution | Total
Number analyzed (Participants) | 42 | 46 | 42 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.22) | 61.7 (9.13) | 60.7 (11.91) | 61.6 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 10 | 23
  Male | 36 | 39 | 32 | 107
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35 | 43 | 37 | 115
  Black or African American | 3 | 2 | 3 | 8
  Asian | 2 | 0 | 2 | 4
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 0 | 1 | 0 | 1
  Hispanic or Latino | 7 | 12 | 9 | 28
  Not Hispanic or Latino | 35 | 34 | 33 | 102
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 46 | 42 | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clearing of Corneal Fluorescein Staining at Week 5 at Week 5
Description: A patient will be considered a success for clearing of corneal fluorescein staining if their fluorescein staining has disappeared
Time Frame: 5 weeks
Population: Full Analysis Set: All patients randomly assigned to receive double-masked study drug, who received at least 1 dose of study drug in the study eye, and who had at least 1 post-baseline assessment for the primary efficacy endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.0002% SJP-0035 Ophthalmic Solution | 0.001% SJP-0035 Ophthalmic Solution
Number analyzed (Participants) | 42 | 45 | 42
Participants | 5 | 7 | 12

ADVERSE EVENTS:
Time Frame: Up to 30 days following final dose (Week 5)
Description: A Treatment-Emergent Adverse Event (TEAE) is defined as any event not present before exposure to study drug, or any event already present that worsens in either intensity or frequency after exposure to study drug.
Arm/Group | Placebo | 0.0002% SJP-0035 Ophthalmic Solution | 0.001% SJP-0035 Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/46 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/46 | 1/42
Other Adverse Events (participants affected / at risk) | 10/42 | 6/46 | 15/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | 0.0002% SJP-0035 Ophthalmic Solution (N=46) | 0.001% SJP-0035 Ophthalmic Solution (N=42)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | 0.0002% SJP-0035 Ophthalmic Solution (N=46) | 0.001% SJP-0035 Ophthalmic Solution (N=42)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival Hyperaemia (Eye disorders) | 2 (4) | 2 (4) | 2 (4)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Retinal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blepharal Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 1 (2) | 0 (0) | 1 (2)
Eye Pain (Eye disorders) | 1 (1) | 0 (0) | 1 (2)
Viral Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Eye Pruritus (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Erythema of Eyelid (Eye disorders) | 0 (0) | 1 (2) | 1 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous Floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Foreign Body Sensation in Eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Viral Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pinguecula (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Trichiasis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival Disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Blood Creatine Phosphokinase (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glare (Eye disorders) | 0 (0) | 0 (0) | 1 (4)
Eye Discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator will not disclose information regarding this clinical investigation, or publish results of the investigation without authorization from Senju Pharmaceuticals Co., Ltd.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT02929823/Prot_SAP_000.pdf